CLINICAL TRIAL: NCT01333215
Title: Etude Des Troubles de l'Inhibition Cognitive Chez le Sujet âgé déprimé Suicidant
Brief Title: Study of Cognitive Inhibition Disorders in Depressed Older Suicide Attempters
Acronym: ETIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Stéphane Richard-Devantoy, Angers University hospital
Other Study IDs: 2010/24
Record Dates: First submitted 2011-04-07; First posted 2011-04-11 (Estimated); Last update posted 2011-04-11 (Estimated); Status verified 2010-12

CONDITIONS: Suicide, Attempted; Cognitive Symptoms
Keywords: Suicide, Attempted; Cognitive Symptoms
MeSH Terms: conditions — Suicide, Attempted; Neurobehavioral Manifestations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group 1: Depressed older suicide non-attempters
- Group 2: Depressed older suicide attempters

SUMMARY:
The purpose of this study is to compare the cognitive inhibition deficit among depressed older suicide attempters compared to depressed older suicide non-attempters.

DETAILED DESCRIPTION:
The main objective consists in examining the association between cognitive inhibition and suicide attempt in depressed older adults (> 65 year old).

ELIGIBILITY:
Inclusion Criteria:

* Age > 65 years old
* Score of Mini-Mental State Examination (MMSE) > 23
* Score of Hamilton Depression Scale >27
* For Group 1 (depressed older suicide non-attempters): No history of suicide attempt
* For Group 2 (depressed older suicide attempters) : History of suicide attempt

Exclusion Criteria:

* Neurological history or medical-surgical affection in the past 3 months.
* Dependence or alcohol abuse.
* Use of neuroleptics

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Patients are recruited during their hospitalisation at Angers University Hospital with respect to the eligibility criteria
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-07 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Cognitive inhibition deficit | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Stephane Richard-Devantoy, Mr., Principal Investigator — Angers University Hospital
Locations (1):
- University Hospital, Angers, France

REFERENCES:
- [Derived] Richard-Devantoy S, Annweiler C, Le Gall D, Garre JB, Olie JP, Beauchet O. Cognitive inhibition in suicidal depressed elderly: a case-control pilot study. J Clin Psychiatry. 2011 Jun;72(6):871-2. doi: 10.4088/JCP.10l06797. No abstract available. PMID 21733483